CLINICAL TRIAL: NCT01907685
Title: An Open Label, Dose Escalation, Safety and Pharmacokinetic Phase 1 Study With AVE8062 Administered as a 30 Minutes Intravenous Infusion Followed by Docetaxel Administered as an 1 Hour Intravenous Infusion 24 Hours-Apart Every 3 Weeks in Patients With Advanced Solid Tumors
Brief Title: Dose Escalation, Safety and Pharmacokinetic Study of AVE8062 Combined With Docetaxel in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD6295; 2005-005027-34 (EudraCT Number)
Record Dates: First submitted 2013-07-15; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Advanced Neoplastic Disease
MeSH Terms: interventions — AC 7700; Docetaxel

ARMS (1):
- AVE8062 / Docetaxel (Experimental): AVE8062 30-minute IV, 11.5 to 42 mg/m2, followed by Docetaxel, 1-hour IV, 75 and 100 mg/m2 in 3-week cycles until disease progression or unacceptable toxicity or study discontinuation criteria
  Interventions: Drug: AVE8062; Drug: Docetaxel

INTERVENTIONS:
Drug: AVE8062 — Pharmaceutical form:Solution for infusion
  Route of administration: Intravenous
  Other Names: Ombrabulin
Drug: Docetaxel — Pharmaceutical form: solution for infusion
  Route of administration: Intravenous
  Other Names: XRP6976

SUMMARY:
Primary Objective:

To determine the dose limiting toxicity (DLT), the maximum administered dose (MAD) and the maximum tolerated dose (MTD) of AVE8062 and docetaxel in combination administered sequentially on D1 & D2 respectively every 3 weeks in patients with advanced solid tumors.

Secondary Objectives:

* To define the overall safety profile of the combination.
* To characterize the pharmacokinetic (PK) profile of AVE8062 and docetaxel when administered in combination.
* To evaluate anti-tumor activity of the combination.
* To evaluate potential predictive biomarkers.

The study includes a tumoral pharmacogenomic sub-study conducted in a subset of sites. The objective to analyse a set of biological biomarkers in order to identify a potential predictive signature of efficacy for AVE8062 in combination with docetaxel.

DETAILED DESCRIPTION:
The duration of study for each patient will include 4-week screening phase prior to first inclusion of study drug, 21-day study treatment cycles, end of treatment visit and follow-up phase. Each patient will be treated until disease progression, unacceptable toxicity or other study discontinuation criteria.

ELIGIBILITY:
Inclusion criteria:

* Advanced neoplastic disease (i.e metastatic or locally advanced disease) for which docetaxel-based regimen therapy is indicated such as breast, non-small cell lung and prostate cancer.
* ECOG performance status of 0 to 1.

Exclusion criteria:

* Concurrent treatment with any other anticancer therapy.
* Patient with locally advanced or metastatic breast cancer who never received adjuvant chemotherapy.
* Brain metastases and carcinomatous leptomeningitis.
* Prior intensive chemotherapy with autologous stem cell rescue.
* Patients who received a high cumulative dose of anthracycline (i.e doxorubicin > 400mg/m2 or epirubicin >750 mg/m2).
* Impaired cardiovascular function.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2006-06; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | 3 weeks (cycle 1)

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | Up to disease progression or unacceptable toxicity or study discontinuation criteria (median treatment of 4 cycles)
Plasma concentration of AVE8062 and its metabolite | Before AVE8062 infusion, immediately prior to the end of AVE8062 infusion, 5, 10, 25, 45 and 60 minutes then 2, 4, 6, 8-10 and 24 hours post AVE8062 infusion (cycle 1)
Plasma concentration of docetaxel | Before docetaxel infusion (corresponding to 24 hours post AVE8062 infusion), 15 minutes before the end of docetaxel infusion, 15 and 45 minutes post docetaxel infusion (cycle 1)
Response evaluation criteria in solid tumors (RECIST) defined objective response | Up to disease progression or unacceptable toxicity or study discontinuation criteria (median treatment of 4 cycles)
Biomarkers expression profile of each patient in order to identify preliminary correlation with antitumor activity of the combination treatment in patients with available pre-treatment biopsy | End of treatment or until disease progression or unacceptable toxicity or study discontinuation criteria

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi

REFERENCES:
- [Derived] Eskens FA, Tresca P, Tosi D, Van Doorn L, Fontaine H, Van der Gaast A, Veyrat-Follet C, Oprea C, Hospitel M, Dieras V. A phase I pharmacokinetic study of the vascular disrupting agent ombrabulin (AVE8062) and docetaxel in advanced solid tumours. Br J Cancer. 2014 Apr 29;110(9):2170-7. doi: 10.1038/bjc.2014.137. Epub 2014 Apr 8. PMID 24714750